CLINICAL TRIAL: NCT02607579
Title: A Randomized, Blinded Study to Compare Exparel and Ropivacaine for Pain Relief Following Total Knee Arthroplasty
Brief Title: Comparing Exparel & Ropivacaine for Pain Relief in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Monmouth Medical Center (Other)
Responsible Party: Principal Investigator, Ryan Plyler, Orthopaedic Surgeon/ Researcher, Monmouth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-045
Record Dates: First submitted 2015-07-27; First posted 2015-11-18 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Ropivacaine (Active Comparator): This group is given an adductor canal block with Ropivacaine which is the previous gold standard medication.
  Interventions: Drug: Ropivacaine
- Exparel (Experimental): This group is given an adductor canal block with Exparel which is believed to last longer and provide a better pain relief post-operatively.
  Interventions: Drug: Exparel

INTERVENTIONS:
Drug: Exparel
  Arms: Exparel
Drug: Ropivacaine
  Arms: Ropivacaine

SUMMARY:
The purpose of this prospective study is to examine the effect of two local anesthetics used in adductor canal blocks, with relation to pain, analgesic consumption, mobility, and pain related interference with activities and hospital length of stay. The two agents are bupivacaine and ropivacaine. The purpose of this trial is to examine the effect of these drugs being used in adductor canal blocks for pain relief, analgesic consumption, mobility, and pain related interference with activities and hospital length of stay.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is associated with intense early postoperative pain. Effective pain management following total knee arthroplasty is imperative to facilitate early ambulation, mobilization and rehabilitation. The postoperative pain regimen should enhance functional recovery in addition to providing efficient analgesia with minimal side effects. To manage postoperative pain effectively, multimodal analgesia including acetaminophen, Toradol, Solu-Medrol, opioids and local anesthetics are used. Periarticular infiltration performed intra-operatively combined with ultrasound guided adductor-canal peripheral nerve blocks are effective in reducing pain following a TKA without causing quadriceps motor block which can impede mobilization. There are no published trials that the investigators could find to date, comparing adductor canal block with a single dose Exparel and adductor canal block with standard ropivacaine.

A liposome is a manufactured spherical lipid vesicle that can be used to slowly release a drug thereby extending its duration of action. Exparel is such a compound that slowly releases bupivacaine. Local anesthetics block the conduction of all excitable tissue in a dose related fashion. The first tissues that are affected are nerves, which make these drugs of choice in neural block. Their local adverse effects include neurovascular manifestations are prolonged numbness, tingling, feeling of "pins and needles" or strange sensations. These effects are reversed with time. There are no additional potential risks or adverse effects due to the procedures or drugs being administered. The procedure is well established and the local anesthetics have a history of long term use in humans.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and up undergoing a total knee replacement with single surgeon. American Society of Anesthesiologists Physical Status Classification Scale (ASA) 1-3.

Exclusion Criteria:

* Allergy to local anesthestic, pre-existing peripheral neuropathy, revision surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Pain relief | Hospital course (approximately 2-3 days)
  The investigators will monitor patient pain scores every 6 hours during the hospital stay based on the Defense and Veterans Pain Rating Scale (DVPRS).

SECONDARY OUTCOMES:
Length of stay | Hospital course (approximately 2-3 days)
  The investigators will compare the length of stay between the two groups.
Post-Operative Range of Motion | Hospital course (approximately 2-3 days)
  The investigators will compare the range of motion between the two groups during the participants' hospital course as measured by the physical therapists on a daily basis.
Post-Operative Distance Walked | Hospital course (approximately 2-3 days)
  The investigators will compare the distance walked between the two groups during the participants' hospital course as measured by the physical therapists on a daily basis.
Amount of Narcotics required | Hospital course (approximately 2-3 days)
  The investigators will monitor the amount of medication taken by participants during the hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Monmouth Medical Center, Long Branch, New Jersey, United States